CLINICAL TRIAL: NCT04039802
Title: Single-stage Bone-anchored Hearing Implant Surgery in the Pediatric Population Using the BHX Implant
Brief Title: Single-stage Surgery Using the BHX Implant
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-5408
Record Dates: First submitted 2019-04-23; First posted 2019-07-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2023-09

CONDITIONS: Hearing Impairment, Conductive; Hearing Impaired Children
Keywords: Single-stage surgery; Bone conduction devices; Pediatric population; Implant loss
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test: In the test group, patients will be scheduled for bone-anchored hearing implant surgery using the single-stage procedure. The implant and abutment will be placed in one surgery
  Interventions: Procedure: Single-stage surgery
- Control: Historical control group, these patients already underwent BAHI insertion using two-stage surgery. The implant and abutment were inserted in two different procedures
  Interventions: Other: Two-stage surgery

INTERVENTIONS:
Procedure: Single-stage surgery — In the test group, patients will be scheduled for bone-anchored hearing implant surgery using the single-stage procedure. The implant and abutment will be placed in one surgery.
  Groups: Test
Other: Two-stage surgery — Two-stage surgery has already been performed, data will therefore be retrospectively collected
  Groups: Control

SUMMARY:
Over the last few decades, the classical two-stage surgical procedure for inserting bone-anchored hearing implants (BAHIs) has been modified in adults into a single-stage procedure. This approach has several advantages since it avoids a second surgical procedure. The single-stage approach is proven to be safe and feasible in adults and is nowadays referred to as the standard surgical technique in adults. Despite favorable outcomes and advantages of the single-stage surgery, most Ear Nose Throat (ENT) surgeons still perform two-stage surgery when inserting BAHI in the pediatric population. Therefore, the aim of this study is to compare implant loss between single-stage BAHI surgery and two-stage BAHI surgery in children aged 4 to 9 years.

DETAILED DESCRIPTION:
General description:

A prospective comparative study with historical control group will be performed.The test group will consist of 22 children aged 4-9 years old who are found to be suitable candidates for treatment with a BAHI (BHX implant and abutment). The control group consists of approximately 50 children, aged 4-9 years old, who already underwent insertion with a wide diameter implant between 2012 and 2018. In the test group, BAHI insertion will be performed using single-stage surgery. Patients in the control group already underwent BAHI insertion using two-stage surgery.

Recruitment and consent:

All children planned for implantation with bone-anchored hearing implants will be screened for inclusion in the present study. Patients who meet the inclusion criteria will be approached for participation by their ENT-specialist, after patients' and parents/caretakers' approval they will be informed and screened for participation by one of the researchers. The study protocol will be discussed with the potential study participant and his/her parents/caretakers by the researcher. The potential study participant and his/her parents/caretakers will be given/sent the Informed Consent Form to read. Potential study participants will be encouraged to discuss the study with family members and personal physician(s) before deciding whether to participate in the study. Patients and their parents/caretakers have 14 days to consider their decision. In order to participate in the study, both parents/caretakers need to sign the informed consent form.

Data handling:

Data captured will be recorded in Castor using electronic Case Report Forms (eCRFs). All data, patient and product related, must be accurately recorded in the eCRF by the delegated site staff. All users of the Castor system have personal, password protected accounts allowing tracking of all data entry in the system. Data management and data cleaning will be performed in the eCRF using the queries function to ensure traceability of all data entry and changes by the assigned data manager. Data including patient identifying information (i.e. name, initials, birth date) will be stored on a secured network drive using a code. Only the investigator who has the code can correlate the data with the patient's name and date of birth. It is the responsibility of the investigator to make sure that patient identification listings with patient code and identity are kept. Raw measurement data and other data such as historical information will be storedin the patient file, since data may be partly acquired and/or evaluated during standard patient care to limit the amount of extra procedures and hospital visits. For data analyses, data will be exported and stored in a digital research environment, separate from the key to the code. After completion of the study data collection and final monitoring visit, the electronic database will be locked and exported to SPSS format, which will be archived for 15 years after completion of the study. The coded study data will be archived separately from the key to the subject code in a secured digital research environment, also for a period of 15 years.

Reporting (severe) adverse events:

The investigator will report the Severe Adverse Events (SAEs) through the web portal ToetsingOnline to the accredited Medical Ethical Committee (METC) that approved the protocol, within 7 days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the investigator has first knowledge of the serious adverse events.

Device deficiency:

Inadequacy of an investigational medical device related to its identity, quality, durability, reliability, safety or performance. This may include malfunctions, use error, or inadequacy in the information supplied by the manufacturer. Device deficiency's will be logged together with an assessment by the investigator and reported to the manufacturer where applicable.

Follow-up of adverse events:

All Adverse Events (AEs) will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist. SAEs need to be reported until the end of study within the Netherlands, as defined in the protocol.

Monitoring and Quality Assurance:

In accordance with the guidelines of the 'Dutch Federation of university medical centers' (NFU) for monitoring of studies with negligible risk, a qualified monitor of another department of the Radboudumc, who is not part of the research team of this study, will be appointed. 28% of informed consents, 10% of inclusion and exclusion criteria (and three subjects who were enrolled first), 10% source data verification, reported SAEs and 10% of participants with regard to missed SAEs will be monitored.

Statistical analysis:

The main analyses will be the comparison between the test group, in which single-stage surgery is performed and the control group undergoing two-stage surgery.

Concerning the primary outcome, the proportions of implant loss in the test and control group will be compared using an exact binominal test and a one tailed confidence interval of 95%.

Secondary outcome measures will be compared between groups using the unpaired t-test (normally distributed data or Mann-Whitney U tests (not normally distributed data) for continuous variables, Mantel Haenszel chi-square test for ordered categorical variables, Fisher's exact test for dichotomous variables and Chi-square test for non-ordered categorical variables. If significant differences are found for baseline variables between the test group and the control group a complementary analysis between the two groups will be performed with adjustment for these variables.

Handling of missing data for secondary and tertiary endpoints (especially applicable for control group data), depends on the reason why this data is missing and on the amount of missing data. Therefore decisions on handling of missing data will be made after all data is collected.

All tests will be performed using a confidence interval of 95% and a significance level of 0.05

ELIGIBILITY:
Inclusion criteria test group:

* Age 4-9 years
* Indication for percutaneous bone-anchored hearing implant surgery with a BI300 implant
* Insertion using the linear incision technique

Inclusion criteria control group:

* Children who underwent implantation of a wide diameter implant using two- stage surgery between 2012 and 2018 at the Radboudumc
* Age 4-9 at the time of surgery
* Linear incision technique was used during surgery

Exclusion Criteria test group:

* Inability to show up at all follow-up visits
* Patients undergoing re-implantation
* Diseases, syndromes or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus.
* Insufficient bone thickness ≤1mm, since conversion to two-stage surgery will be advocated

Exclusion Criteria control group

* Follow-up duration less than 1 year.
* Diseases, syndromes or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus (at moment of implantation)

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 4 to 9 years old who are planned for treatment with a BAHI (BI300 implant) are considered candidates for the study. They will be approached for participation in the trial after they have chosen a Cochlear sound processor after thorough clinical and audiological testing and counseling. These patients are selected from a tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Implant loss | 1 year
  The number of lost implants

SECONDARY OUTCOMES:
Soft-tissue status according to Holgers scale | 1 year
  The Holgers scale is a worldwide used soft tissue assessment scale for percutaneous implants for BCDs. The degree of soft tissue reactions is classified as follows27:
  0 = No irritation
  1. = Slight redness
  2. = Red and slightly moist tissue
  3. = Reddish and moist; sometimes granulation tissue
  4. = Removal of skin-penetrating implant necessary due to infection R = Removal of implant for reasons not related to skin problems Holgers score of 2 or higher is considered to be an adverse skin reaction
Soft-tissue status according to IPS | 1 year
  The IPS scale is a relatively new consistent, uniform, and easy assessment scale for both percutaneous and transcutaneous implants for BCDs.28 For percutaneous implants, the IPS-scale comprising three parts: inflammation, pain, and skin height, with higher scores reflecting more severe complication. It assesses the following characteristics:
  1. Inflammation:
     * Skin Integrity (intact = 0 / not intact = 1)
     * Erythema (none = 0 / present = 1)
     * Edema (none = 0 / present = 1)
     * Granulation tissue formation (none = 0/ present = 1)
  2. Pain:
     * None = 0
     * Present, but no increase during manipulation abutment AND <6 wks present = 1
     * Present, and increase during manipulation abutment AND/OR >6 wks present = 2
  3. Skin height:
     * Normal = 0
     * Increased, but able to couple sound processor = 1
     * Above rim abutment/unable to couple sound processor =2 An IPS score equal to or higher than I1P1S0/I2P0S0/I0P2S0/I0P0S2
Time to loading | through study completion, an average of 1 year
  Time from first surgery until loading of sound processor
Duration of surgery | through study completion, an average of 1 year
  In test group duration of single-stage surgery. In the control group duration of first and second surgery together

CONTACTS AND LOCATIONS:
Overall Officials: Hol, dr, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saliba I, Froehlich P, Bouhabel S. One-stage vs. two-stage BAHA implantation in a pediatric population. Int J Pediatr Otorhinolaryngol. 2012 Dec;76(12):1814-8. doi: 10.1016/j.ijporl.2012.09.007. Epub 2012 Sep 23. PMID 23010336
- [Background] Kohan D, Morris LG, Romo T 3rd. Single-stage BAHA implantation in adults and children: is it safe? Otolaryngol Head Neck Surg. 2008 May;138(5):662-6. doi: 10.1016/j.otohns.2007.12.019. PMID 18439475
- [Background] Ali S, Hadoura L, Carmichael A, Geddes NK. Bone-anchored hearing aid A single-stage procedure in children. Int J Pediatr Otorhinolaryngol. 2009 Aug;73(8):1076-9. doi: 10.1016/j.ijporl.2009.03.028. Epub 2009 May 26. PMID 19473711
- [Background] Marsella P, Scorpecci A, D'Eredita R, Della Volpe A, Malerba P. Stability of osseointegrated bone conduction systems in children: a pilot study. Otol Neurotol. 2012 Jul;33(5):797-803. doi: 10.1097/MAO.0b013e318255dd73. PMID 22643446
- [Background] de Wolf MJ, Hol MK, Huygen PL, Mylanus EA, Cremers CW. Nijmegen results with application of a bone-anchored hearing aid in children: simplified surgical technique. Ann Otol Rhinol Laryngol. 2008 Nov;117(11):805-14. doi: 10.1177/000348940811701103. PMID 19102125
- [Background] Mazita A, Fazlina WH, Abdullah A, Goh BS, Saim L. Hearing rehabilitation in congenital canal atresia. Singapore Med J. 2009 Nov;50(11):1072-6. PMID 19960162